CLINICAL TRIAL: NCT03058068
Title: A Phase I, Randomized and Placebo-controlled Trial to Evaluate the Safety, Tolerability, and Potential Efficacy of Allogeneic Human MesenchymAl Stem Cells Infusion in Patients With Cystic Fibrosis - HAPI
Brief Title: Human MesenchymAl Stem Cells Infusion in Patients With Cystic Fibrosis
Acronym: HAPI
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI left the institution
Sponsor: Joshua M Hare (Other)
Responsible Party: Sponsor-Investigator, Joshua M Hare, Sponsor, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20160140
Record Dates: First submitted 2017-02-06; First posted 2017-02-20 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: 1. Safety run-in phase will have 3 subjects with 2 treatment groups
  2. Randomized phase will have 15 subjects with 3 treatment groups
Who Masked: Participant, Investigator
Masking Description: Masking will apply to the randomized phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Safety Run-In: Treatment 1 Allo-hMSCs (Experimental): Treatment 1: 1 subject will receive a single administration of allogeneic MSCs: 20 x 10^6 MSCs (20 million) cells delivered via peripheral intravenous infusion.
  Interventions: Biological: Allo-hMSCs
- Safety Run-In: Treatment 2 Allo-hMSCs (Experimental): 2 subjects will receive a single administration of allogeneic MSCs: 100 x 10^6 MSCs (100 million) cells delivered via peripheral intravenous infusion.
  Interventions: Biological: Allo-hMSCs
- Randomized: Cohort 1 Allo-hMSCs (Experimental): Cohort 1 (5 subjects): 20 million MSCs A single peripheral intravenous infusion of 20 x 10^6 MSCs (20 million cells) will be administered to each subject.
  Interventions: Biological: Allo-hMSCs
- Randomized: Cohort 2 Allo-hMSCs (Experimental): Cohort 2 (5 subjects): 100 million MSCs A single peripheral intravenous infusion of 100 x 10^6 MSCs (100 million cells) will be administered to each subject.
  Interventions: Biological: Allo-hMSCs
- Randomized: Cohort 3 Allo-hMSCs (Placebo Comparator): Cohort 3 (5 subjects): Placebo A single peripheral intravenous infusion of placebo (PlasmaLyte A containing 1% HSA) will be administered to each subject.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Allo-hMSCs — 1 peripheral intravenous infusion of allogeneic human mesenchymal stem cells (hMSCs)
  Other Names: Stem cells
  Arms: Randomized: Cohort 1 Allo-hMSCs; Randomized: Cohort 2 Allo-hMSCs; Safety Run-In: Treatment 1 Allo-hMSCs; Safety Run-In: Treatment 2 Allo-hMSCs
Biological: Placebo — 1 peripheral intravenous infusion
  Arms: Randomized: Cohort 3 Allo-hMSCs

SUMMARY:
A Safety Run-In will be followed by a Double-Blinded Randomized Phase. All subjects shall meet the inclusion/exclusion criteria, and will be evaluated prior to the scheduled infusion to establish baseline.

There will be 3 subjects in the safety run-in phase and 15 subjects in the double-blinded phase.

DETAILED DESCRIPTION:
Primary objective is to demonstrate the safety of Mesenchymal Stem Cells (MSCs) intravenously administered to subjects with cystic fibrosis.

Secondary Objective is to explore if MSCs can improve the symptoms of cystic fibrosis, including lung function, the rate of pulmonary exacerbation, systemic and local inflammation and symptom-related quality of life.

The Safety Run-In will be performed to evaluate the safety of MSC infusion into subjects with cystic fibrosis. 3 subjects will participate and they will receive a single administration of allogeneic MSCs given through intravenous infusion.

In the randomized phase the subjects will be randomized at a ratio of 1:1:1 into 3 cohorts to receive infusions. There will be a total of 15 subjects in 3 cohorts.

The total duration for each subject after infusion is 12 months, plus up to an additional 2 months for the Screening and Baseline Visits. Approximately 9 visits in total.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent.
* Be 20 - 45 years of age at the time of signing the Informed Consent Form.
* Have a confirmed diagnosis of cystic fibrosis as defined by two or more clinical features of cystic fibrosis (CF), including by the 1997 CF

Consensus criteria (NIH Consensus Statement, 1997):

One or more accompanying clinical features consistent with Cystic fibrosis, and at least one of the following:

1. Documented sweat chloride test ≥ 60 mEq/L by quantitative pilocarpine iontophoresis or,
2. Abnormal nasal transepithelial potential difference (NPD) test or,
3. Two well-characterized, disease-causing genetic mutations in the CF transmembrane conductance regulator (CFTR) gene on different alleles

   * FEV1 at screening visit between 25% and 80% of predicted values for age, sex, and height taken 4 hours or more after last dose of short-acting bronchodilators (β-agonists and/or anticholinergics). The predicted values will be calculated according to National Health and Nutrition Examination Survey (NHANES).
   * Total bilirubin below 1.9 mg/dL.
   * Non-smoker for the past 60 days (2 months) prior to screening Visit 1 and less than a 5 pack-year lifetime history of smoking
   * Stable regimen of CF medications and chest physiotherapy for the 28 days prior to screening, and no anticipated need for changes during the study period for the immediate future, at least 4 weeks post infusion.
   * Clinically stable for at least 4 weeks with no evidence of new or acute respiratory symptoms, excluding symptoms of allergic (perennial or seasonal) or non-allergic rhinitis.
   * Patients should be on a stable medication regimen as determined by their Cystic fibrosis physician. Allowable medications include:

     * Inhaled medications (bronchodilators, steroids, pulmozyme, hypertonic saline and inhaled antibiotics to suppress chronic infections including tobramycin, amikacin, colistin, aztreonam lysine)
     * Chronic azithromycin use (three times weekly)
     * Vitamin supplementation
     * Pancreatic enzymes
     * CFTR potentiator and/or corrector (ivacaftor and lumacaftor)

Exclusion Criteria:

All subjects enrolled in this trial must not:

* Be unable to perform any of the assessments required for endpoint analysis.
* Use systemic corticosteroids (≥5 mg of prednisone per day).
* Have been on intravenous or oral antibiotics within the last 4 weeks
* Have a clinical history of malignancy within 5 years (i.e., subjects with prior malignancy must be disease free for 5 years), except curatively- treated basal cell carcinoma, squamous cell carcinoma, melanoma in situ or cervical carcinoma, if recurrence occurs.
* Have congestive heart failure (NYHA Class III or IV).
* Have severe pulmonary hypertension with a right ventricle systolic pressure (RVSP) >50 mmHg as estimated by echocardiography
* Have chronic kidney disease Stage 4 or 5.
* Have a non-pulmonary condition that limits lifespan to ≤1 year.
* Have clinically significant autoimmune disease (e.g., rheumatoid arthritis, systemic lupus erythematosus (SLE), or inflammatory bowel disease).
* Have HIV, AIDS, or other immunodeficiency.
* Test positive for hepatitis B HsAg, viremic hepatitis C, HIV1, HIV2, HTLV-I, HTLV-II, syphilis, and West Nile Virus.
* Have a resting blood oxygen saturation of <93% (measured by pulse oximetry).
* Have documented current substance and/or alcohol abuse.
* Be a current user of tobacco products.
* Have a known hypersensitivity to dimethyl sulfoxide (DMSO).
* Have had a recent (within prior 3 months) trauma or surgery.
* Be an organ transplant recipient.
* Be actively listed (or expected to be listed) for transplant of any organ other than for a lung transplant.
* Have any clinically important abnormal screening laboratory values, including but not limited to:

  * hemoglobin <12.1 g/dL (females) or <13.6 g/dL (males).
  * white blood cell count < 3000/mm3.
  * platelets < 150,000/mm3.
  * International normalized ratio (INR) ˃ 1.5 not due to a reversible cause (i.e. Coumadin).
  * aspartate transaminase, alanine transaminase, or alkaline phosphatase ˃ 2 times upper limit of normal.
* Have a sitting or resting systolic blood pressure >180 mm Hg or diastolic blood pressure >110 mm Hg at Screening.
* Have any serious comorbid illness or any other condition that, in the opinion of the Investigator, may compromise the safety or compliance of the patient or preclude successful completion of the study, or that may compromise the validity of the study.
* Be a female who is pregnant, nursing, or of childbearing potential while not practicing effective contraception (female patients must undergo a blood or urine pregnancy test at screening and prior to infusion). Females who are in childbearing age must agree to practice a highly effective form of contraception throughout the study. Highly effective forms of contraception with a low failure rate include barrier methods, oral contraception or depot contraceptives (unless on Orkambi), an intrauterine device, implantable devices.
* Be currently participating in an investigational therapeutic or device trial, or have participated in an investigational therapeutic or device trial within the previous 30 days, or participate in any other clinical trial for the duration of the time that the subject actively participates in this trial.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of any treatment-emergent serious adverse event (TE-SAE) | 30 days after infusion
  Incidence of any treatment-emergent serious adverse event (TE-SAE), defined as one or more of the following untoward medical occurrences happening within the first 30 days after infusion.

SECONDARY OUTCOMES:
Change in Symptoms for pulmonary function test | baseline to 12 months
  examining post-infusion changes from baseline between the MSC and Placebo Cohorts in terms of:
  • Resting pulmonary function tests (PFTs) assessed via spirometry: forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1), FEV1 to FVC ratio, and forced expiratory flow between 25 - 75% of VC (FEF25-75) measured in adherence to American Thoracic Society/European Respiratory Society guidelines.
Change in Symptoms 6-minute walk test | baseline to 12 months
  examining post-infusion changes from baseline between the MSC and Placebo Cohorts in terms of:
  • 6-minute walk test (6MWT).
Change in Symptoms of body mass index | baseline to 12 months
  examining post-infusion changes from baseline between the MSC and Placebo Cohorts in terms of:
  • Changes in body mass index
Change in Rate of pulmonary exacerbations | baseline to 12 months
  examining post-infusion changes from baseline between the MSC and Placebo Cohorts in terms of:
  * Incidence of investigator-defined pulmonary exacerbation: events meeting the modified Fuchs' criteria (at least 4 of 12 signs and symptoms with or without intravenous or oral antibiotic treatment).
  * Semi-quantitative sputum cultures (change in colony forming units)
  * Procalcitonin serum levels
Change in Local and Systemic Inflammation in inflammatory markers | baseline to 12 months
  examining post-infusion changes from baseline between the MSC and Placebo Cohorts in terms of:
  • Serum Inflammatory markers (CBC with differential, TNFα, C-reactive protein, Interleukin-1, Interleukin-6, D-dimer, Fibrinogen).
Change in Local and Systemic Inflammation for sputum inflammatory markers | baseline to 12 months
  examining post-infusion changes from baseline between the MSC and Placebo Cohorts in terms of:
  • Sputum inflammatory markers
Change in Local and Systemic Inflammation related to quality of life | baseline to 12 months
  examining post-infusion changes from baseline between the MSC and Placebo Cohorts in terms of:
  • Symptom Related Quality of Life
Change in Local and Systemic Inflammation via the short form-36 | baseline to 12 months
  examining post-infusion changes from baseline between the MSC and Placebo Cohorts in terms of:
  • Physical activity via the short form-36 questionnaires.
Change in Local and Systemic Inflammation via the PHQ-9 Questionnaire | baseline to 12 months
  examining post-infusion changes from baseline between the MSC and Placebo Cohorts in terms of: • Subject quality of life (QOL) assessments via:
  - Patient Health Questionnaire-9 (PHQ-9) for depression screening
Change in Local and Systemic Inflammation via the CFQ-R Questionnaire | baseline to 12 months
  examining post-infusion changes from baseline between the MSC and Placebo Cohorts in terms of: • Subject quality of life (QOL) assessments via:
  - Cystic Fibrosis Questionnaire-Revised (CFQ-R)
Change in Local and Systemic Inflammation via the GAD-7 Questionnaire | baseline to 12 months
  examining post-infusion changes from baseline between the MSC and Placebo Cohorts in terms of: • Subject quality of life (QOL) assessments via:
  - Generalized anxiety disorder 7 (GAD-7)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias A Salathe, MD, Principal Investigator — ISCI / University of Miami / Division of Pulmonary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Interdisciplinary stem cell institute (ISCI) at the University of Miami — http://isci.med.miami.edu